CLINICAL TRIAL: NCT02843269
Title: Multiple-component Workplace FRamed Intervention to Decrease Occupational Muscle Pain - FRIDOM. Background, Design and Conceptual Model of a Cluster Randomized Double-blinded Controlled Study Among Female Health Care Workers
Brief Title: Multiple-component Workplace FRamed Intervention to Decrease Occupational Muscle Pain - FRIDOM
Acronym: FRIDOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Jeanette Reffstrup Christensen, PHD, University of Southern Denmark
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: S-20130157
Record Dates: First submitted 2016-06-23; First posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-07

CONDITIONS: Neck Pain; Shoulder Pain; Lifestyle
Keywords: RCT; Multi-component intervention; Health personnel; Physical exercise training
MeSH Terms: conditions — Neck Pain; Shoulder Pain

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Multi-component lifestyle intervention 1 (Active Comparator): A multi-component intervention consisting of Intelligent Physical Exercise training (IPET), Dietary Advice and Weight loss (DAW) and Cognitive Behavioral Therapy (CBT)
  Interventions: Behavioral: Multi-component lifestyle intervention
- Multi-component lifestyle intervention 2 (Active Comparator): A multi-component intervention consisting of Intelligent Physical Exercise training (IPET), Dietary Advice and Weight loss (DAW) and Cognitive Behavioral Therapy (CBT)
  Interventions: Behavioral: Multi-component lifestyle intervention
- Multi-component lifestyle intervention 3 (Active Comparator): A multi-component intervention consisting of Intelligent Physical Exercise training (IPET), Dietary Advice and Weight loss (DAW) and Cognitive Behavioral Therapy (CBT)
  Interventions: Behavioral: Multi-component lifestyle intervention

INTERVENTIONS:
Behavioral: Multi-component lifestyle intervention — The exact same intervention was given to the three Stepped-wedge groups - but each of the three groups were started up three months apart. The waiting groups served as control groups. Thus, the intervention were for all three groups a multi-component intervention consisting of Intelligent Physical Exercise training (IPET), Dietary Advice and Weight loss (DAW) and Cognitive Behavioral Therapy (CBT)

SUMMARY:
Several RCT studies have aimed to reduce either musculoskeletal disorders, sickness presenteeism, sickness absenteeism or a combination of these among females with high physical work demands. These studies have provided evidence that workplace health promotion (WHP) interventions are effective, but long-term effects are still uncertain. These studies either lack to succeed in maintaining intervention effects or lack to document if effects are maintained past a one-year period. FRIDOM (FRamed Intervention to Decrease Occupational Muscle pain) is a WHP program among health care workers. A job group characterized by having high physical work demands, musculoskeletal disorders, high sickness presenteeism - and absenteeism.

FRIDOM aimed to reduce neck and shoulder pain and secondary to reduce sickness presenteeism and sickness absenteeism. An other secondary aim was to decrease lifestyle-diseases such as other musculoskeletal disorders as well as metabolic-, and cardiovascular disorders - and to maintain participation to regular physical exercise training, after a one year intervention period. The entire concept was tailored to a population of female health care workers. This was done through a multi-component intervention including 1) intelligent physical exercise training (IPET), dietary advice and weight loss (DAW) and cognitive behavioural training (CBT).

DETAILED DESCRIPTION:
The FRIDOM program was composed of four parts: 1) A planning phase according to intervention mapping principles, 2) a feasibility study to reveal issues of implementation and intervention content, 3) a randomized controlled trial (RCT) , and 4) a maintenance period. Below these components are further detailed.

Intervention mapping and time frame The main focus of the intervention was on sustainable behavioural life-style changes, therefore, a key point was a detailed planning of all phases to ease the final maintenance of the introduced health enhancing activities after the 12 months supervised intervention.

The FRIDOM-Feasibility study To prepare and facilitate the FRIDOM-RCT study a feasibility study was conducted which served several purposes. Before the intervention in the feasibility study was initiated, all eligible employees were asked to fill out a screening questionnaire and participate in a baseline-screening-test. To allow for subsequent adjustment of the intervention content and mode of practical implementation, the feasibility study was timed ahead of the RCT study, according to the same principal schedule as the RCT.

The FRIDOM-RCT study The FRIDOM-RCT was implemented as a cluster RCT with a "stepped wedge" design. Content of the intervention had to be given repeatedly, and it was an important step to avoid changes in intervention delivery to the successive cohorts.

The FRIDOM-Maintenance Besides the primary and secondary goals, it was a long term goal to implement the intervention elements as permanent activities at the workplace, maintained beyond the one-year intervention period. Therefore, the activities offered at the workplace should include not only baseline consenters, but also gradually involve new employees and employees returning to work.

Study population The FRIDOM program was offered to the entire elderly care section in a medium size municipality in Jutland, Denmark. All eligible personnel at the entire elderly care section was invited to participate in the project to optimize motivation to comply with the intervention.

Recruitment Procedure A necessary number of meetings were held to reach all eligible participants. Prior to the meetings, written information was distributed to the employees in a short information pamphlet. Managers supplied employees, who did not attend the information meeting with written information and a screening questionnaire.

The FRIDOM-Feasibility study The feasibility study included both health care workers, working in centers for elderly people and retirement homes and employees working in the elderly´s private home in both day, evening and night shifts.

The FRIDOM-RCT The RCT participants were individually allocated to a team according to the following criteria for minimizing variation within a team: 1) Geographical location of the workplace, 2) working at center/home care facilities or in the elderlies private home, and 3) day or evening/night shifts. To maximize motivation by social bonding with colleagues within a team, close relations with colleagues were taken into consideration. In order to minimize contamination between clusters, priority was given to minimize variation in geographical location within a cluster.

Intervention content The one-hour weekly multi-component intervention consisted of a combination of intelligent physical exercise training (IPET) including Power Breaks, dietary advice and weight loss (DAW) and cognitive behavioral therapy (CBT).

IPET The principles for IPET were that the exercise training was adjusted to 1) occupational physical exposure, 2) physical capacity, 3) health status and 4) motivations and barriers.

The physical exercise consisted of two elements: strength training exercises with elastic band as resistance (Power Breaks) and aerobic exercises. The aerobic exercises were inspired by the protocol developed in a previously workplace study.

DAW All participants were guided to ensure a healthy diet and prevent weight gain by adjusting courses according to the Danish Dietary recommendations. For each individual the resting metabolism was calculated, based on gender, age and weight and multiplied by a Physical Activity Level factor of 1.8 to estimate the daily energy requirement. ~1.000 calories were subtracted from the estimated daily energy requirements and the resulting value was used as individual calorie prescription.

CBT The CBT training was developed in a previous research project by Christensen. The CBT was provided as group discussions and followed a specifically tailored guideline, containing exercises such as pro-and-con schemes and homework between each session. To support the aim of participant adherence to workplace physical exercise and regular leisure time physical exercise training, motivational initiatives based upon Self-Determination Theory were included.

Instructors Due to Danish legislation, all employees were entitled to six weeks vacation. Thus, weekly training sessions were only carried out in 46 weeks and were all supervised with instructors.

Outcome measures Outcome measures were collected in four different categories: (Category 1) data drawn from workplace registrations, (category 2) questionnaires, (category 3) physiological tests and (category 4) adherence. Besides the physical tests, the physiological tests included blood samples of blood sucker, cholesterol and triglyceride. Category 1-4 tests were collected on all participants, in either the FRIDOM-feasibility or the FRIDOM-RCT study. At some time points, a full packages of each category were collected (Large test), while at other time points, only a subsets were collected (Mini test). Besides the Large tests and the Mini tests, a screening test was initially conducted.

Workplace registrations (1) Information about age, sex, job seniority, weekly working hours, work shift, care center or home care, job type and educational level were gathered from the workplaces own registration on their employees. Sickness absenteeism were retrieved from a local database maintained by the executive director at the workplace.

Questionnaire (2) The FRIDOM program consisted of three different questionnaires. 1) A Large questionnaire given at baseline and followed-up after one year within each RCT-cluster, 2) a Mini questionnaire to be completed every third months, and finally 3) a Screening questionnaire distributed before randomization. The Large questionnaire involved lifestyle behaviour and health, dietary intake, physical activity during leisure time, self-rated health and Stress-Energy Scale, SF-36, physical resources with five items: aerobic fitness, strength, endurance, flexibility and balance/coordination, readiness to change, Cohens Perceived Stress Scale, chronic diseases, Standardized Nordic Questionnaires of musculoskeletal symptoms last seven days and pain intensity on a numeric rank box scale, general self-efficacy, Tampa Scale of Kinesiophobia, Work ability Scale, perceived physical exertion, productivity by a single item in the World Health Organization Health and Work Performance Questionnaire (HPQ) and Quantity and Quality of work.

The Mini questionnaire every third months consisted of eight questions, included the Standardized Nordic Questionnaires for the analysis of musculoskeletal symptoms last seven days and pain intensity, physical capacity, balance/coordination, readiness to change and general self-efficacy.

The Screening questionnaire consisted of a subset of items from the Large questionnaire. The purpose was to evaluating reach of the intervention within the RE-AIM framework. Pain was measured by Standardized Nordic Questionnaires for the analysis of musculoskeletal symptoms last 12 months.

Physiological tests (3) The FRIDOM program included three different test-batteries. A large test-battery measured at baseline and after one year, a Mini test every third months and a Screening test before randomization. All participants were tested with a Large test at baseline and after one year of intervention. The large test lasted one hour and consisted of anthropometrical, health-related and physical capacity measures such as height, body weight, body fat, waist circumference, blood pressure, aerobic fitness, isometric maximal voluntary strength in hands, shoulder elevation, back flexion and extension force.

The Mini tests lasted 15 minutes and included: blood pressure, body weight, BMI, body fat, waist circumference, and balance test.

The Screening test lasted 3 minutes and included information's on weight, BMI and body fat.

Adherence (4) Participation in the 46 weekly multi-component training offered at the workplace were registered by the instructors. Performance of daily five minutes exercise with elastic bands (Power Breaks), color of the Thera band, and number of windings (1-3) were reported in a training diary.

Additional measures in a nested subsample Diurnal measurements consisting of physical activity and electrocardiogram were performed on a random subset of participants. Physical activity was subsequently quantified as time in sitting, standing and walking using custom build software.

Electrocardiogram for estimation of heart rate and heart rate variability was recorded using e-Patch data loggers initialized with gender and age using the commercial software Hasimed. During the diurnal measurements, participants were asked to follow their normal every-day schedule life and to note in a paper diary, working hours, sleeping and waking time, and if any of the monitors were removed before scheduled.

Statistics Analysis of outcome were performed both on the entire population and on the health care target population. The primary outcome measure was questionnaire based self-reported duration and intensity of neck pain with all other outcome measures considered secondary outcomes. For the Feasibility study the pre-post test were analyzed using paired t-test and repeated measures. For the RCT difference between the three clusters at baseline were to be tested with Pearson´s x² for distribution in sex, education, current smoking status and the dichotomized parameter for musculoskeletal symptoms in neck, shoulders, upper- and lower back. All other parameters were to be tested with a Student´s t-test. Changes over the 3 months intervention periods were compared with the changes over the corresponding 3 months control periods in an ANCOVA analysis in accordance to the intention-to-treat principle, i.e. all randomized participants were included in the analyses with missing values substituted with carried forward or backwards measured variables. Clusters, age and the investigated value at baseline were included as covariates. All results were given as mean (SD). P<0.05 were considered statistically significant. SPSS statistics 23 was used for the statistical analysis.

In order to account for the combined effect within and between subjects and repeated measurements on the same subject, linear mixed effects models were used. Additionally, likelihood ratio tests was used to compare the models with and without a covariance structure. Analyses were based on the intention to treat principle including all eligible participants without imputations since mixed effects models inherently account for missing values.

Sample size for the RCT part was estimated using the method described by Woertman & colleagues for sample size calculation. The study was powered to detect a between-groups mean difference in the primary endpoint of 1 point in pain intensity, which has been considered a relevant change in the workplace context in terms of risk of sickness absence. The variance was set to 2.0 based on results from a Danish study within a similar population, α to 0.05, power to 0.8, and an intra-cluster correlation coefficient to 0.05 in the three steps. The calculation showed that 82 participants in total were needed and with a dropout rate of up to 50% it was planned to recruit at least 160 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Participants should be employed at the elderly care department at a Danish municipality (Sydjurs).
2. Working at least 15 hours per week.
3. Permanently employed, or
4. Have at least 12 months of work left before retirement.

Exclusion Criteria:

1. Long-term sick listed.
2. Pregnancy, or
3. Working at a rehabilitation center, as these employees do not have work tasks within elderly care

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 219 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Neck pain intensity as assessed by a 10 point Visual Analogue Scale | 12 months follow-up
Shoulder pain intensity as assessed by a 10 point Visual Analogue Scale | 12 months follow-up

SECONDARY OUTCOMES:
Risk factors for lifestyle diseases - Blood pressure with an electronic blood pressure monitoring device | Baseline, 1, 3 and 5 years
  From baseline to 1, 3 and 5 years follow-up with an electronic blood pressure monitoring device (Artsana CS 410)
Risk factors for lifestyle diseases - Body fat using a bio impedance device | Baseline, 1, 3 and 5 years
  From baseline to 1, 3 and 5 years follow-up using a bio impedance device (TANITA SC-330)
Risk factors for lifestyle diseases - Waist circumference using an ergonomic circumference measuring tape | Baseline, 1, 3 and 5 years
  From baseline to 1, 3 and 5 years follow-up using an ergonomic circumference measuring tape (Seco 203 Girth measuring tape)
Risk factors for lifestyle diseases - Aerobic fitness with the Wattmax test | Baseline, 1, 3 and 5 years
  From baseline to 1, 3 and 5 years follow-up measured with the Wattmax test using a Monark E327 bicycle ergometer and a pulse belt
Sickness absence retrieved from a local database | Baseline, 1, 3 and 5 years
  sickness absence were retrieved from a local database maintained by the executive director at the workplace, from 1 year before intervention start to 1, 3 and 5 years follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette R Christensen, PHD, Principal Investigator — University of Southern Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ilvig PM, Bredahl TVG, Justesen JB, Jones D, Lundgaard JB, Sogaard K, Christensen JR. Attendance barriers experienced by female health care workers voluntarily participating in a multi-component health promotion programme at the workplace. BMC Public Health. 2018 Dec 4;18(1):1340. doi: 10.1186/s12889-018-6254-3. PMID 30514352
- [Derived] Christensen JR, Bredahl TV, Hadrevi J, Sjogaard G, Sogaard K. Background, design and conceptual model of the cluster randomized multiple-component workplace study: FRamed Intervention to Decrease Occupational Muscle pain - "FRIDOM". BMC Public Health. 2016 Oct 24;16(1):1116. doi: 10.1186/s12889-016-3758-6. PMID 27776506